CLINICAL TRIAL: NCT00752479
Title: Mesenchymal Stem Cells Under Basiliximab/Low Dose RATG to Induce Renal Transplant Tolerance
Acronym: MSC-KTX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Necessity of major revision of the protocol
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MSC KTX; 2009-012350-20 (EudraCT Number)
Record Dates: First submitted 2008-07-23; First posted 2008-09-15 (Estimated); Last update posted 2023-12-04 (Actual); Status verified 2015-04

CONDITIONS: Kidney Transplant
Keywords: living; related
MeSH Terms: interventions — Basiliximab; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Mesenchymal stem cells infusion, Basiliximab,Methylprednisolone,RATG ,Cyclosporine ,Mycophenolate mofetil
- 2 (Active Comparator)
  Interventions: Drug: Basiliximab, Methylprednisolone,RATG,Cyclosporine,Mycophenolate mofetil

INTERVENTIONS:
Biological: Mesenchymal stem cells infusion, Basiliximab,Methylprednisolone,RATG ,Cyclosporine ,Mycophenolate mofetil — Cell therapy
  Mesenchymal cells infusion.
  Induction therapy:
  Basiliximab (20 mg i.v.day 0 and day 4 post-tx). Low dose RATG (0.5 mg/kg/day i.v. day 0-6 post-tx). Methylprednisolone (500 mg to 25 mg from day 0 to 6 post-tx. Then stop).
  Maintenance therapy:
  Cyclosporine (from day 0: dose according to target trough blood level). Mycophenolate mofetil (750 mg b.i.d. from day 1 post-tx).
  Arms: 1
Drug: Basiliximab, Methylprednisolone,RATG,Cyclosporine,Mycophenolate mofetil — Routine immunosuppressive therapy
  Induction therapy:
  Basiliximab (20 mg i.v.day 0 and day 4 post-tx). Low dose RATG (0.5 mg/kg/day i.v. day 0-6 post-tx). Methylprednisolone (500 mg to 25 mg from day 0 to 6 post-tx. Then stop).
  Maintenance therapy:
  Cyclosporine (from day 0: dose according to target trough blood level). Mycophenolate mofetil (750 mg b.i.d. from day 1 post-tx).
  Arms: 2

SUMMARY:
This a pilot, explorative study to define the safety and biological/mechanistic effect of the systemic intravenous infusion of syngeneic ex-vivo expanded MSCs in living-related kidney transplant recipients (one or two HLA haplotype mismatches) under basiliximab/low-dose RATG induction therapy and maintenance immunosuppressive drugs with the ultimate objective to test the feasibility of safely achieving graft tolerance in a subsequent efficacy pilot study.

Specific objectives To compare changes in the immunophenotype and ex-vivo T-cell functional tests from samples of peripheral blood and measurement in the urine of messenger RNA for FoxP3,in kidney transplant recipients given or not syngeneic (from the recipient) MSC infusion under basiliximab/low-dose RATG induction therapy and maintenance immunosuppressive treatment with low-dose cyclosporine (CsA) plus low-dose mycophenolate mofetil (MMF).

This will assess at different time up to 12 months post transplant. In addition the safety profile of MSC infusion will be investigated. We have planned to start with the safety and biological/mechanistic study in 6 living-related kidney transplant recipients. Three patients will receive ex-vivo expanded syngeneic MSC infusion (2x106 MSCs per kilogram body weight) at the time of kidney transplant, and 3 additional patients no cells (controls), both under the cover of induction therapy with basiliximab and low-dose RATG, and maintenance immunosuppression with low-dose CsA and MMF. Randomization to MSC or no cell infusion will be performed at the time the recipient will sign the informed consent to participate to the study.

Should this biological/mechanistic ex vivo studies document that MSC infusion allows the development of an immune microenvironment permissive to graft tolerance, a pilot efficacy study to achieve operational tolerance after complete withdrawal of maintenance immunosuppressive therapy will follow.

In this additional pilot explorative efficacy study all consecutive patients will be included and followed until the first episode of rejection (if any) will occur or 29 consecutive patients have successfully withdrawn the immunosuppressive therapy. This has been estimated according to the Simon's two-stage minimax design.

DETAILED DESCRIPTION:
INTRODUCTION In organ transplantation the immunosuppressive drugs have dramatically improved the life of transplant recipients over the past 30 years, but two notable problems remain:drug-associated toxicities, and failure of these drugs to prevent chronic graft dysfunction and extend long-term graft survival. Given these circumstances, the scientific discussion is dominated by designing effective ways to induce transplantation tolerance. 'Transplantation tolerance' describes a state in which a donor is 'accepted' without chronic immunosuppressive therapy, while the remainder of the immune system is left intact. Thus, lack of a pathogenic response to the alloantigen is specific, and the recipient is capable of responding to potentially pathogenic microorganisms and malignancies. There is abundant evidence for active immunoregulatory mechanisms, which may operate to maintain transplant tolerance.

The problems of immunosuppressive drug toxicity could be alleviated by induction of immune tolerance.Over the last 25 years, several strategies have been used successfully to induce transplantation tolerance. Each of these has been validated in at least one rodent model, with varying degrees of success upon extension to large animals, including nonhuman primates. Very small minorities of patients, who discontinue their immunosuppression, provide rare examples of clinical transplantation tolerance. To this purpose, mesenchymal stem cell (MSC) infusion could represent a novel tolerogenic cell therapy in kidney transplantation.

Human bone marrow stem cells, more recently referred to as MSCs, are multipotential cells that reside within the bone marrow and can differentiate into various components of the marrow microenvironment, in addition to supporting growth of hematopoietic progenitors.There is also evidence that MSCs escape the immune system, and therefore could be infused into an allogeneic host without being rejected and without requirement of conditioning regimens. Moreover, they exert an immunoregulatory activity, although the exact mechanism of action is unknown. On this line, evidence is available that MSC inhibit naïve T cells and lock dendritic cells (DC) into a semi-mature state, thereby favoring peripheral tolerance. It should be also pointed out that experimental in vitro evidence has shown that mouse MSCs inhibit the response of memory antigen-specific T cells to their cognate peptide. We expect that, in kidney transplant recipients, MSC infusion would allow inhibition of alloantigen-specific memory T cell response contributing to long-term graft survival. Moreover in vitro studies have documented that the CD4+CD25+ T regulatory cell population increased significantly in MLR when human MSCs were present compared to controls without MSCs. These findings suggest that MSC may modulate T cell response even through a regulatory mechanism. Furthermore an immunosuppressive effect of MSCs in vivo has been shown in a baboon model, in which infusion of ex-vivo expanded matched donor or third-party MSCs delayed the time to rejection of histoincompatible skin graft. The immunomodulatory function of MSCs has been also documented in preliminary in vivo studies in humans, where cell infusion did exert preventive effects on the development of acute and chronic GVHD. Thus, although no data so far are available in human kidney transplantation, we expect that peri-transplant intravenous infusion of syngeneic ex-vivo expanded MSCs under peripheral T-cell depletion/blockade with basiliximab and low dose RATG (as induction therapy) and the cover of low dose maintenance immunosuppressive drugs would allow to safety achieving graft tolerance in living-related kidney transplant recipients. This could be through inhibition of both naïve and memory T cells, and promotion of development and activation of regulatory T cells, eventually leading to indefinite graft survival.

Up to now there is no clinical study that MSC infusion has an immunomodulatory effect in patients undergoing kidney transplant. Nevertheless, there are clinical data on the effectiveness and safety of MSC infusion in other diseases/conditions.

The general aim of the present study is to test a cell therapy with syngeneic ex vivo expanded MSC as a strategy to induce tolerance in living-related kidney transplant recipients. MSC will be prepared accordingly to established protocols, starting from bone marrow explants of living-related recipients obtained 3-4 months before kidney transplant. From these samples, MSC will be expanded in vitro and used for the present study in patients undergoing kidney transplantation.

AIMS AND STUDY DESIGN This a pilot, explorative study to define the safety and biological/mechanistic effect of the systemic intravenous infusion of syngeneic ex-vivo expanded MSCs in living-related kidney transplant recipients (one or two HLA haplotype mismatches) under basiliximab/low-dose RATG induction therapy and maintenance immunosuppressive drugs with the ultimate objective to test the feasibility of safely achieving graft tolerance in a subsequent efficacy pilot study. Indeed, to complement the research with a clinical portion that document operational tolerance, a pilot efficacy study of safely achieving kidney graft tolerance after complete withdrawal of maintenance immunosuppressive therapy will follow pending on the fact that the results of biological/mechanistic tests will document that MSC infusion allows the development of an immune microenvironment permissive to graft tolerance.

Specific objectives To compare changes in the immunophenotype and ex-vivo T-cell functional tests from samples of peripheral blood and measurement in the urine of messenger RNA for FoxP3,in kidney transplant recipients given or not syngeneic (from the recipient) MSC infusion under basiliximab/low-dose RATG induction therapy and maintenance immunosuppressive treatment with low-dose cyclosporine (CsA) plus low-dose mycophenolate mofetil (MMF).

In particular, at different time up to 12 months post transplant, the plan is the following:

Immunophenotyping

1. To assess the effect of the treatment on absolute and percent count of circulating CD4+, CD8+ T cells (and the CD4/CD8 ratio), B cells and NK cells.
2. To examine whether changes in circulating naïve and memory T cell count may occur (CD45RA/CD45RO).
3. To characterize the emergence in the circulation of T cell subpopulations with immunoregulatory phenotype (CD4+CD25highFOXP3+; CD8+CD28-, CD3-CD56bright).

Lymphocyte functional assays

1. To detect whether donor-specific hyporesponsiveness develops post-operatively by monitoring T cell activation in response to alloantigen stimulation by mixed lymphocyte reaction (MLR), by ELISPOT assay for IFN-gamma and by cell-mediated lympholysis (CML).
2. To determine whether T cell deletion/anergy develops by repeating T cell stimulation in MLR and in IFN-gamma ELISPOT assay in the presence of high doses of IL-2.
3. To monitor the regulatory properties of T cells circulating in the peripheral blood by in vitro proliferative assay, in particular of CD4+CD25high, CD8+CD28- T cells, and CD56bright NK cells.

Urinary FOXP3 messenger RNA

a)To evaluate whether measurement in urinary cells of mRNA level for FoxP3, a functional factor for regulatory T lymphocytes, may provide insight into the immunologic events within the renal allograft.

In addition the safety profile of MSC infusion will be investigated.

Should this biological/mechanistic ex vivo studies document that MSC infusion allows the development of an immune microenvironment permissive to graft tolerance, a pilot efficacy study to achieve operational tolerance after complete withdrawal of maintenance immunosuppressive therapy will follow. The criteria to document the development of a pro-tolerogenic microenvironment (at 12 months post-kidney transplant) are the followings:

* Percentage of inhibition of memory T cell response (by IFN-gamma ELISPOT) and/or naïve T cell response (by MLR) versus donor antigens higher than 15-20% in patients receiving peri-transplant MSC infusion as compared to patients receiving the immunosuppressive therapy alone, in the context of normal immune responses versus third party antigens, mitogens (PHA) and recall antigens (mumps, pertussis).

and

* Induction of donor-reactive T cell anergy in a percentage higher than 15-20% in patients receiving peri-transplant MSC infusion as compared to those given the immunosuppressive therapy alone (evaluated by addition of high dose IL-2 in ELISPOT assay) or
* Appearance in the peripheral blood of regulatory T cells in a percentage higher than 80% in patients receiving peri-transplant MSC infusion as compared to patients receiving the immunosuppressive therapy alone and reversal of the inhibition of donor-specific immune response (evaluated by depletion of specific regulatory cells in ELISPOT and/or MLR assays) in a percentage higher than 50% in MSC-treated as compared with non MSC-treated patients.

We have planned to start with the safety and biological/mechanistic study in 6 living-related kidney transplant recipients. Three patients will receive ex-vivo expanded syngeneic MSC infusion at the time of kidney transplant, and 3 additional patients no cells (controls), both under the cover of induction therapy with basiliximab and low-dose RATG, and maintenance immunosuppression with low-dose CsA and MMF. Randomization to MSC or no cell infusion will be performed at the time the recipient will sign the informed consent to participate to the study. This will be when the patients fulfill all the criteria to enter the waiting list for kidney transplant from living donor.

The first patient will receive a single i.v infusion of syngeneic MSC (2x106 MSCs per kilogram body weight). If the procedure is safe and no major adverse events related to the i.v cell infusion will occur within the first month (early peri-infusion side effects, severe infections possibly due to over-immunosuppression), the second patients will be enrolled. Should the procedure be safe also in this case, the third kidney transplant patient will be enrolled and undergo syngeneic MSC infusion.

To complement this research with a clinical portion that document operational tolerance, a pilot efficacy study of safely achieving kidney graft tolerance after complete withdrawal of maintenance immunosuppressive therapy will follow pending on the fact that the results of biological/mechanistic tests (at 12 months post-transplant) will document that MSC infusion allows the development of an immune microenvironment permissive to graft tolerance, as higher inhibition of donor specific memory T cells and/or higher generation of alloantigen-specific regulatory T cells than the drug immunosuppressive treatment alone.

In this additional pilot explorative efficacy study all consecutive patients will be included and followed until the first episode of rejection (if any) will occur or 29 consecutive patients have successfully withdrawn the immunosuppressive therapy. This has been estimated according to the Simon's two-stage minimax design.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Aged 18 or older
* Non-HLA identical with the donor (one or two haplotype mismatches)
* First kidney transplant
* Capable of understanding the purpose and risk of the study
* Written informed consent

Exclusion Criteria:

* MSC donor positive for HIV-1, HIV-2, HBV, HCV, Syphilis.
* Specific contraindication to MSC infusion
* Any clinical relevant condition that might affect study participation and/or study results
* Pregnant women and nursing mothers
* Unwillingness or inability to follow study protocol in the investigator's opinion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assessing the percentage of inhibition of memory T cell response and/or naive T cell response, the induction of donor-reactive T cell anergy and the appearance in the peripheral blood of regulatory T cells. | at 12 months post-kidney transplant

SECONDARY OUTCOMES:
Safety parameters related to MSC infusion, graft function, graft rejection | at 12 months post-kidney transplant

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, MD, Study Chair — Department of Immunology and Clinical Transplantation / Mario Negri Institute for Pharmacological Research and Ospedali Riuniti BG; Norberto Perico, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research, Ranica BG; Marina Noris, CH Ph, Principal Investigator — Mario Negri Institute for Pharmacological Research, Ranica BG; Martino Introna, MD, Principal Investigator — Cell and Gene therapy Laboratory "G. Lanzani" BG; Alessandro Rambaldi, MD, Principal Investigator — Hematology Unit - Ospedali Riuniti BG
Locations (1):
- Nephrology Unit, Bergamo, BG, Italy

REFERENCES:
- [Derived] Perico N, Casiraghi F, Todeschini M, Cortinovis M, Gotti E, Portalupi V, Mister M, Gaspari F, Villa A, Fiori S, Introna M, Longhi E, Remuzzi G. Long-Term Clinical and Immunological Profile of Kidney Transplant Patients Given Mesenchymal Stromal Cell Immunotherapy. Front Immunol. 2018 Jun 14;9:1359. doi: 10.3389/fimmu.2018.01359. eCollection 2018. PMID 29963053
- [Derived] Perico N, Casiraghi F, Gotti E, Introna M, Todeschini M, Cavinato RA, Capelli C, Rambaldi A, Cassis P, Rizzo P, Cortinovis M, Noris M, Remuzzi G. Mesenchymal stromal cells and kidney transplantation: pretransplant infusion protects from graft dysfunction while fostering immunoregulation. Transpl Int. 2013 Sep;26(9):867-78. doi: 10.1111/tri.12132. Epub 2013 Jun 6. PMID 23738760
- [Derived] Perico N, Casiraghi F, Introna M, Gotti E, Todeschini M, Cavinato RA, Capelli C, Rambaldi A, Cassis P, Rizzo P, Cortinovis M, Marasa M, Golay J, Noris M, Remuzzi G. Autologous mesenchymal stromal cells and kidney transplantation: a pilot study of safety and clinical feasibility. Clin J Am Soc Nephrol. 2011 Feb;6(2):412-22. doi: 10.2215/CJN.04950610. Epub 2010 Oct 7. PMID 20930086